CLINICAL TRIAL: NCT01307995
Title: Observational Study to Evaluate the Reduced Incretin Effect Observed in Patients With GDM in Relation to Reversibility After a Delivery.
Brief Title: The Incretin Effect in Patients With Gestational Diabetes Mellitus
Status: Completed | Type: Observational
Sponsor: Medical University of Lodz (Other)
Collaborators: University of Copenhagen (Other)
Responsible Party: Marcin Kosinski, Diabetology and Metabolic Diseases Departament
Other Study IDs: GDM-INK
Record Dates: First submitted 2011-03-02; First posted 2011-03-03 (Estimated); Last update posted 2011-03-03 (Estimated); Status verified 2011-01

CONDITIONS: Gestational Diabetes
Keywords: GDM; incretin effect; gestation; reversibility
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Observational Model: Case-Crossover
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- GDM: Patients with Gestational Diabetes Mellitus found during pregnancy by means of 75g OGTT
- NGT: Pregnant patients with normal glucose tolerance as observed in 75g OGTT

SUMMARY:
The aim of this study is to evaluate the reduced incretin effect observed in patients with T2DM in relation to reversibility. The incretin effect will be measured by means of OGTT and iIVGTT in 12 women with GDM during pregnancy (third trimester), and again 2-3 months post partum. It is anticipated that the incretin effect in patients with GDM is reduced - like in patients with other forms of DM. The investigators estimate that approximately 90 % of the patients with GDM re-establish a NGT 2-3 months post partum. This particular group of patients provides a unique possibility for demonstrating the reversibility of the reduced incretin effect in relation to optimal glycaemic control.

ELIGIBILITY:
Inclusion Criteria:

* age above 18 years old
* GDM diagnosed according to WHO guidelines (GDM group) or ruled out by OGTT 75g (Control group)

Exclusion Criteria:

* Previous diagnosis of DM
* Positive GAD-65-autoantibodies and/or positive islet cell autoantibodies (ICA)
* Affected biochemical liver parameters (ALAT > 2 times normal upper range)
* Affected biochemical kidney parameters (se-creatinine > 130 µM)
* Treatment with medicine interacting with insulin secretion (e.g. steroids)
* Treatment with medicine that can not be paused for 16 hours

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Pregnant women above the age of 18 years with GDM) (Controls: pregnant women above the age of 18 years with NGT)
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2007-04; Primary Completion 2009-12 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Katarzyna Cypryk, MD, PhD, Asoc. Prof., Study Director — Medical University Lodz; Tina Vilsbøll, MD, DMSc, Study Director — University of Copenhagen; Marcin Kosiński, MD, PhD, Principal Investigator — Medical University Lodz
Locations (1):
- Departament of Diabetology and Metabolic Diseases, Polish Mothers Research Hospital, Lodz, Poland